CLINICAL TRIAL: NCT03404609
Title: Rapid Non-Invasive Brain Stimulation for OCD (oTMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43421
Record Dates: First submitted 2018-01-13; First posted 2018-01-19 (Actual); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: OCD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Accelerated course of modified continuous theta-burst stimulation (cTBSmod) (Experimental): Participants received 5 consecutive days of accelerated cTBSmod to the right frontal pole. Each cTBSmod session was comprised of 1800 pulses, delivered in a continuous train of 600 bursts. Each burst contained 3 pulses at 30 Hz, repeated at 6 Hz. Ten sessions were applied per day (18,000 pulses/day, hourly) (90,000 total pulses) using a Magventure Magpro X100. Stimulation was delivered at 90% resting motor threshold (depth corrected). Localite Neuronavigation System was used to position the TMS coil over the individualized stimulation target.
  Interventions: Device: MagPro X100 by MagVenture

INTERVENTIONS:
Device: MagPro X100 by MagVenture — Participants received 5 consecutive days of accelerated cTBSmod to the right frontal pole. Each cTBSmod session was comprised of 1800 pulses, delivered in a continuous train of 600 bursts. Each burst contained 3 pulses at 30 Hz, repeated at 6 Hz. Ten sessions were applied per day (18,000 pulses/day, hourly) (90,000 total pulses) using a Magventure Magpro X100. Stimulation was delivered at 90% resting motor threshold (depth corrected). Localite Neuronavigation System was used to position the TMS coil over the individualized stimulation target.

SUMMARY:
The purpose of this study is to understand how cortical stimulation affects Obsessive-Compulsive Disorder (OCD) symptoms.

DETAILED DESCRIPTION:
Obsessive-Compulsive Disorder (OCD) is a chronic and disabling disorder that costs the economy over $2 billion annually and represents a significant public health problem. This study aims to understand how cortical stimulation affects Obsessive-Compulsive Disorder

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Primary diagnosis of OCD
* Sufficient severity of OCD symptoms
* Capacity to provide informed consent

Exclusion Criteria:

* Psychiatric or medical conditions or medications that make participation unsafe
* Pregnant or nursing females
* Previous exposure to TMS or ECT
* History of any implanted device or psychosurgery
* Presence of metallic device or dental braces

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Rodriguez, MD, PhD, Principal Investigator — Stanford University; Nolan Williams, MD, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Result] Williams NR, Sudheimer KD, Cole EJ, Varias AD, Goldstein-Piekarski AN, Stetz P, Lombardi A, Filippou-Frye M, van Roessel P, Anderson K, McCarthy EA, Wright B, Sandhu T, Menon S, Jo B, Koran L, Williams LM, Rodriguez CI. Accelerated neuromodulation therapy for Obsessive-Compulsive Disorder. Brain Stimul. 2021 Mar-Apr;14(2):435-437. doi: 10.1016/j.brs.2021.02.013. Epub 2021 Feb 23. No abstract available. PMID 33631349
- See also: Rodriguez Lab — http://med.stanford.edu/rodriguezlab.html

RESULTS

PARTICIPANT FLOW:
Groups:
- rTMS: Participants in the rTMS group will receive MagPro X100 by MagVenture (Active) cortical stimulation condition.
  MagPro X100 by MagVenture: Participants in the rTMS group will receive MagPro X100 by MagVenture cortical stimulation condition.
Period: Overall Study
Arm/Group | rTMS
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | rTMS
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Met and Exceeded Response Criteria of Yale-Brown Obsessive-Compulsive Scale.
Description: Patients given YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response was defined as at least a 35% reduction on the YBOCS.
Time Frame: Baseline and up to two weeks
Measure: Count of Participants; unit: Participants
Arm/Group | rTMS
Number analyzed (Participants) | 7
Participants | 4

ADVERSE EVENTS:
Time Frame: Baseline and through study completion (e.g., up to approximately 4 weeks)
Arm/Group | rTMS
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS (N=7)
Fatigue (Nervous system disorders) | 3 (3)
headache (Nervous system disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
This pilot study provides preliminary evidence of the safety, feasibility, and efficacy of a 5-day individualized, accelerated, high-dose, cTBSmod protocol for treatment-refractory OCD. Controlled trials are needed to test these promising findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03404609/Prot_SAP_001.pdf